CLINICAL TRIAL: NCT01696747
Title: GpR 2: Continuation of the NIDDK Gastroparesis Registry for the Characterization and Clinical Course of Gastroparesis Patients
Brief Title: Gastroparesis Registry 2
Acronym: GpR2
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: GpCRC-GpR 2-5; U01DK073974 (NIH); U01DK073975 (NIH); U01DK073983 (NIH); U01DK073985 (NIH); U01DK074007 (NIH); U01DK074008 (NIH)
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Gastroparesis; Diabetic Gastroparesis; Idiopathic Gastroparesis
Keywords: gastroparesis; idiopathic gastroparesis; diabetic gastroparesis; post-Nissen gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma serum DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Diabetic: participants with a primary etiology of diabetic gastroparesis
- Idiopathic: participants with a primary etiology of idiopathic gastroparesis
- Post-Nissen: participants with a primary etiology of post-Nissen fundoplication gastroparesis

SUMMARY:
To expand a registry of patients for the study of the epidemiology, etiology, and degree of morbidity associated with gastroparesis.

DETAILED DESCRIPTION:
The Gastroparesis Registry 2 (GpR 2) will enroll new patients and patients from the initial NIDDK Gastroparesis Clinical Research Consortium Gastroparesis Registry (GpR) of gastroparesis patients which was initiated in February 2007 and completed in March 2011.

To continue to follow and expand the data collections of a well-characterized cohort to further define the natural history and clinical course of gastroparesis.

To provide a reliable source for recruitment of well-characterized patients with gastroparesis for therapeutic clinical trials, pathophysiological, molecular, histopathologic, or other ancillary studies. These subsequent clinical trials or ancillary studies will be conducted under separate study protocols with separate consent processes.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis of at least 12 weeks duration (do not have to be contiguous) with varying degrees of nausea, vomiting, early satiety, post-prandial fullness, and/or abdominal pain
* An etiology of either diabetic, idiopathic, or post-Nissen fundoplication gastroparesis
* Gastric emptying scintigraphy of solids and liquids test using 4 hours Egg Beaters® protocol within the last 6 months with either:

  * Abnormal gastric emptying rate defined as an abnormal 2 hour (>60% retention) and/or 4 hour (>10% retention) result based on a 4-hour scintigraphic low fat Egg Beaters® gastric emptying study performed at a GpCRC clinical center.
  * Patients with a normal gastric emptying rate but with symptoms of gastroparesis may be enrolled and classified as possible gastroparesis or gastroparesis-like with normal gastric emptying
* Age at least 18 years at initial screening visit
* Upper endoscopy results within last 2 years

Exclusion Criteria:

* Inability to comply with or complete the gastric emptying scintigraphy test (including allergy to eggs)
* Presence of other conditions that could explain the patient's symptoms:
* Pyloric or intestinal obstruction as determined by endoscopy, upper GI series or abdominal CT scan
* Active inflammatory bowel disease
* Known eosinophilic gastroenteritis
* Primary neurological conditions that could cause nausea and/or vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
* Acute liver failure
* Advanced liver disease (Child's B or C; a Child-Pugh-Turcotte (CPT) score of ≥7 )
* Acute renal failure
* Chronic renal failure (serum creatinine >3 mg/dL) and/or on hemodialysis or peritoneal dialysis
* Total or subtotal (near complete) gastric resection, esophagogastrostomy, gastrojejunostomy, or gastric bypass. Note: patients with prior fundoplication will be eligible for enrollment.
* Any other plausible structural or metabolic cause
* Any other condition, which in the opinion of the investigator would interfere with study requirements
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with gastroparesis and delayed gastric emptying. These patients can have either diabetic, idiopathic, or post-Nissen fundoplication gastroparesis. In addition, patients with symptoms similar to gastroparesis, but with normal gastric emptying will be enrolled as a reference group.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hamilton, MD, MPH, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (6):
- United States (6):
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital-Digestive Healthcare Center, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared at end of funding

REFERENCES:
- [Derived] Parkman HP, Van Natta ML, Maurer AH, Koch KL, Grover M, Malik Z, Sarosiek I, Abell TL, Bulat R, Kuo B, Shulman RJ, Farrugia G, Miriel L, Tonascia J, Hamilton F, Pasricha PJ, McCallum RW. Postprandial symptoms in patients with symptoms of gastroparesis: roles of gastric emptying and accommodation. Am J Physiol Gastrointest Liver Physiol. 2022 Jul 1;323(1):G44-G59. doi: 10.1152/ajpgi.00278.2021. Epub 2022 May 3. PMID 35502871
- [Derived] Parkman HP, Van Natta ML, Makol A, Grover M, McCallum RW, Malik Z, Koch KL, Sarosiek I, Kuo B, Shulman RJ, Farrugia G, Miriel L, Tonascia J, Hamilton F, Pasricha PJ, Abell TL; NIDDK Gastroparesis Clinical Research Consortium. Prevalence and clinical correlates of antinuclear antibody in patients with gastroparesis. Neurogastroenterol Motil. 2022 May;34(5):e14270. doi: 10.1111/nmo.14270. Epub 2021 Oct 1. PMID 34595805
- [Derived] Sarosiek I, Van Natta M, Parkman HP, Abell T, Koch KL, Kuo B, Shulman RJ, Farrugia G, Grover M, Hamilton FA, Pasricha PJ, Yates KP, Miriel L, Wilson L, Yamada G, Tonascia J, McCallum RW; National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Gastroparesis Clinical Research Consortium (GpCRC). Effect of Domperidone Therapy on Gastroparesis Symptoms: Results of a Dynamic Cohort Study by NIDDK Gastroparesis Consortium. Clin Gastroenterol Hepatol. 2022 Mar;20(3):e452-e464. doi: 10.1016/j.cgh.2021.05.063. Epub 2021 Jun 2. PMID 34089855
- [Derived] Pasricha PJ, Grover M, Yates KP, Abell TL, Bernard CE, Koch KL, McCallum RW, Sarosiek I, Kuo B, Bulat R, Chen J, Shulman RJ, Lee L, Tonascia J, Miriel LA, Hamilton F, Farrugia G, Parkman HP; National Institute of Diabetes and Digestive and Kidney Diseases/National Institutes of Health Gastroparesis Clinical Research Consortium. Functional Dyspepsia and Gastroparesis in Tertiary Care are Interchangeable Syndromes With Common Clinical and Pathologic Features. Gastroenterology. 2021 May;160(6):2006-2017. doi: 10.1053/j.gastro.2021.01.230. Epub 2021 Feb 3. PMID 33548234
- [Derived] Parkman HP, Wilson LA, Yates KP, Koch KL, Abell TL, McCallum RW, Sarosiek I, Kuo B, Malik Z, Schey R, Shulman RJ, Grover M, Farrugia G, Miriel L, Tonascia J, Hamilton F, Pasricha PJ; NIDDK/NIH Clinical Gastroparesis Consortium. Factors that contribute to the impairment of quality of life in gastroparesis. Neurogastroenterol Motil. 2021 Aug;33(8):e14087. doi: 10.1111/nmo.14087. Epub 2021 Jan 25. PMID 33493377
- [Derived] Parkman HP, Sharkey E, McCallum RW, Hasler WL, Koch KL, Sarosiek I, Abell TL, Kuo B, Shulman RJ, Grover M, Farrugia G, Schey R, Tonascia J, Hamilton F, Pasricha PJ; NIH/NIDDK Gastroparesis Consortium. Constipation in Patients With Symptoms of Gastroparesis: Analysis of Symptoms and Gastrointestinal Transit. Clin Gastroenterol Hepatol. 2022 Mar;20(3):546-558.e5. doi: 10.1016/j.cgh.2020.10.045. Epub 2020 Oct 28. PMID 33130007
- [Derived] Parkman HP, Van Natta M, Yamada G, Grover M, McCallum RW, Sarosiek I, Farrugia G, Koch KL, Abell TL, Kuo B, Miriel L, Tonascia J, Hamilton F, Pasricha PJ. Body weight in patients with idiopathic gastroparesis. Neurogastroenterol Motil. 2021 Feb;33(2):e13974. doi: 10.1111/nmo.13974. Epub 2020 Sep 15. PMID 32930463
- [Derived] Parkman HP, Sharkey EP, Nguyen LA, Yates KP, Abell TL, Hasler WL, Snape W, Clarke J, Schey R, Koch KL, Kuo B, McCallum RW, Sarosiek I, Grover M, Farrugia G, Tonascia J, Pasricha PJ; Frank A. Hamilton for the NIH Gastroparesis Consortium. Marijuana Use in Patients with Symptoms of Gastroparesis: Prevalence, Patient Characteristics, and Perceived Benefit. Dig Dis Sci. 2020 Aug;65(8):2311-2320. doi: 10.1007/s10620-019-05963-2. Epub 2019 Nov 22. PMID 31758430
- [Derived] Parkman HP, Wilson LA, Hasler WL, McCallum RW, Sarosiek I, Koch KL, Abell TL, Schey R, Kuo B, Snape WJ, Nguyen L, Farrugia G, Grover M, Clarke J, Miriel L, Tonascia J, Hamilton F, Pasricha PJ. Abdominal Pain in Patients with Gastroparesis: Associations with Gastroparesis Symptoms, Etiology of Gastroparesis, Gastric Emptying, Somatization, and Quality of Life. Dig Dis Sci. 2019 Aug;64(8):2242-2255. doi: 10.1007/s10620-019-05522-9. Epub 2019 Mar 9. PMID 30852767
- [Derived] Parkman HP, Yamada G, Van Natta ML, Yates K, Hasler WL, Sarosiek I, Grover M, Schey R, Abell TL, Koch KL, Kuo B, Clarke J, Farrugia G, Nguyen L, Snape WJ, Miriel L, Tonascia J, Hamilton F, Pasricha PJ, McCallum RW. Ethnic, Racial, and Sex Differences in Etiology, Symptoms, Treatment, and Symptom Outcomes of Patients With Gastroparesis. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1489-1499.e8. doi: 10.1016/j.cgh.2018.10.050. Epub 2018 Nov 4. PMID 30404035
- [Derived] Siraj ES, Homko C, Wilson LA, May P, Rao AD, Calles J, Farrugia G, Hasler WL, Koch KL, Nguyen L, Snape WJ, Abell TL, Sarosiek I, McCallum RW, Pasricha PJ, Clarke J, Tonascia J, Hamilton F, Parkman HP. Islet Cell Associated Autoantibodies and C-Peptide Levels in Patients with Diabetes and Symptoms of Gastroparesis. Front Endocrinol (Lausanne). 2018 Feb 13;9:32. doi: 10.3389/fendo.2018.00032. eCollection 2018. PMID 29487566
- [Derived] Orthey P, Yu D, Van Natta ML, Ramsey FV, Diaz JR, Bennett PA, Iagaru AH, Fragomeni RS, McCallum RW, Sarosiek I, Hasler WL, Farrugia G, Grover M, Koch KL, Nguyen L, Snape WJ, Abell TL, Pasricha PJ, Tonascia J, Hamilton F, Parkman HP, Maurer AH; NIH Gastroparesis Consortium. Intragastric Meal Distribution During Gastric Emptying Scintigraphy for Assessment of Fundic Accommodation: Correlation with Symptoms of Gastroparesis. J Nucl Med. 2018 Apr;59(4):691-697. doi: 10.2967/jnumed.117.197053. Epub 2017 Sep 28. PMID 28970332
- [Derived] Parkman HP, Hallinan EK, Hasler WL, Farrugia G, Koch KL, Nguyen L, Snape WJ, Abell TL, McCallum RW, Sarosiek I, Pasricha PJ, Clarke J, Miriel L, Tonascia J, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Early satiety and postprandial fullness in gastroparesis correlate with gastroparesis severity, gastric emptying, and water load testing. Neurogastroenterol Motil. 2017 Apr;29(4):10.1111/nmo.12981. doi: 10.1111/nmo.12981. Epub 2016 Oct 25. PMID 27781342
- See also: Gastroparesis Clinical Research Consortium — https://jhuccs1.us/gpcrc/